CLINICAL TRIAL: NCT01047410
Title: ACtive Care After Transplantation, a Lifestyle Intervention in Renal Transplant Recipients
Brief Title: ACtive Care After Transplantation, the ACT Study
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Kidney Foundation (Other); Innovation Fund of the Dutch Medical Insurance Companies (Unknown)
Responsible Party: Principal Investigator, Eva Corpeleijn, Dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METc 2014/190
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Post-transplant Weight Gain; Kidney Transplant; Metabolic Syndrome
Keywords: physical exercise training; quality of life; exercise capacity; skeletal muscle strength; physical activity level; costeffectiveness; renal transplantation; hemodialysis; peritoneal dialysis; diet
MeSH Terms: conditions — Metabolic Syndrome | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: 3-arm randomized controlled trial
Masking Description: Outcomes assessors are blinded if possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Patients assigned to the usual care group receive the standard medical care (usual care) during the 15 months lasting study period. Physical training does not form a part of the usual care of renal transplant and dialysis patients. After randomisation, patients assigned to the usual care group receive the advice to meet the 'Nederlandse Norm Gezond Bewegen (NNGB), i.e. the advice to perform 30 minutes of moderately intense physical activity at at least five but preferably all days of the week.
- Exercise intervention (Experimental): The exercise intervention in this group is identical to the exercise-only group. Patients assigned to the exercise intervention participate in a 12 weeks lasting, intensive, standardized and supervised physical training program which consists of a combination of endurance and strength training. After completion of the training program, patients receive an individual sport- and physical activity advice and lifestyle coaching.
  Interventions: Other: Exercise intervention
- Exercise intervention and dietary advice (Experimental): The exercise intervention in this group is identical to the exercise-only group. The nutritional intervention runs throughout the entire 15 month intervention. The nutritional intervention aims to critically discuss pre-transplantation nutritional habits, and to set goals for healthier, better quality nutrition to prevent over eating and weight gain. These goals are set together with the subject to facilitate an autonomy supportive coaching climate.During the dietary consults, special attention goes out to saturated fat intake, whole-wheat and high fibre foods, fruit and vegetable intake, dietary salt consumption, and the use of energy-rich beverages such as soda, dairy drinks and fruit juices.
  Interventions: Other: Exercise intervention; Other: Exercise intervention and dietary advice

INTERVENTIONS:
Other: Exercise intervention — Patients assigned to the exercise intervention participate in a 12 weeks lasting, intensive, standardized and supervised physical training program which consists of a combination of endurance and strength training. After completion of the training program, patients receive an individual sport- and physical activity advice and lifestyle coaching.
  Arms: Exercise intervention; Exercise intervention and dietary advice
Other: Exercise intervention and dietary advice — The exercise intervention in this group is identical to the exercise-only group. The nutritional intervention runs throughout the entire 15 month intervention. The nutritional intervention aims to critically discuss pre-transplantation nutritional habits, and to set goals for healthier, better quality nutrition to prevent over eating and weight gain. These goals are set together with the subject to facilitate an autonomy supportive coaching climate.During the dietary consults, special attention goes out to saturated fat intake, whole-wheat and high fibre foods, fruit and vegetable intake, dietary salt consumption, and the use of energy-rich beverages such as soda, dairy drinks and fruit juices.
  Arms: Exercise intervention and dietary advice

SUMMARY:
The aim of the present study is to compare the outcomes of standard care to the effects of exercise alone, and exercise combined with nutrition counseling, on post-transplantation weight gain and quality of life in renal transplant recipients (RTR). The primary outcome is subdomain physical functioning of quality of life, (SF-36 PFS).

Secondary outcomes include other evaluations of quality of life (SF-36, KDQOL-SF, EQ-5D), objective measures of physical functioning (aerobic capacity and muscle strength), level of physical activity, gain in adiposity (body fat percentage by bio-electrical impedance assessment, BMI, waist circumference), and cardiometabolic risk factors (blood pressure, lipids, glucose metabolism). Additionally it is planned to study data on renal function, medical history, medication, psychological factors (motivation, kinesiophobia, coping style), nutrition knowledge, nutrition intake, nutrition status, fatigue, work participation, process evaluation and cost-effectiveness.

DETAILED DESCRIPTION:
Patient and graft survival in the first year after renal transplantation have improved substantially over the last decade, but long-term graft loss and patient mortality have remained high. It is increasingly recognized that the alarmingly poor cardio-metabolic risk profile in renal transplant recipients (RTR) plays a main role in long-term outcome. Improvement of long-term outcome will require specific efforts to improve cardio-metabolic profile and its complications. Importantly, the substantial increase in body weight and body fat that occurs after transplantation is a major trigger for the poor cardiometabolic profile in the RTR, including post-transplant diabetes and metabolic syndrome.

The increase in body weight is mostly fat tissue and typically around 9-10 kg. Most of this weight gain (~90%) occurs in the first year after transplantation. Recent data indicate that steroid avoidance could not prevent this early increase in adiposity. This warrants specific focus on lifestyle factors, i.e diet and physical activity. In the UMCG RTR cohort we found that a lack of physical activity was related to a worse cardiometabolic profile and was an independent predictor of mortality. Moreover, the substantial increase in fat massweight gain was strongly related to low physical activity, high intake of energy-dense drinks, low consumption of vegetables, to increased plasma triglycerides and the metabolic syndrome. The intake of salt and saturated fat was high and fibre intake was low, indicating dietary habits that deviate substantially from recommendations for a healthy diet. Thus, both physical activity and dietary habits are important targets for lifestyle intervention in RTR.

Lasting improvements in lifestyle are notoriously difficult to obtain, but in recent years substantial intervention expertise has been developed in other high risk groups including prediabetes. It is now established that for long term purposes, prevention of excessive weight gain is more effective than treatment of weight excess. Since in RTR most of the weight is gained in the first year after transplantation, prevention is a very promising approach. Moreover, data in prediabetes suggest that combined intervention targeting both diet and physical activity may be particularly effective to this purpose.

Therefore, our aim is to investigate the effects on quality of life by a combined diet-and-physical activity program in RTR in the first year after transplantation.

This randomized controlled intervention study will use a combined diet-and-physical activity approach. After hospital discharge for transplantation, 219 patients will be randomized to three either a control groups: one group, who will receive standard care, one group will be exposed to a 3-month exercise program followed by individual counselling and one group will be exposed to the exercise program + dietary or to intervention followed by individual counselling. The individual counselling is to consolidate the achieved improvements in diet and physical activity and will be provided until 15 months after inclusion. This counselling is based on theories of behavioural change and motivational interviewing. Daily physical activity is evaluated with a pedometer and dietary habits by questionnaires and food records.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Informed Consent;
* >1 year after transplantation
* Medical approvement for participation in the study by the nephrologist.

Exclusion Criteria:

* Psychopathology;
* Severe cognitive disorders;
* Negative advice of the nephrologist and/or cardiologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-10; Primary Completion 2017-08-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Quality of life - Physical Functioning Score | baseline, 12 weeks, 6 months and 15 months
  The subdomain 'Physical Functioning' of Quality of Life (SF36 questionnaire)

SECONDARY OUTCOMES:
Quality of Life Scores | baseline, 12 weeks, 6 months and 15 months
  Physical and Mental scores of the Quality of Life SF36 questionnaire
Physical functioning | baseline, 12 weeks, 6 months and 15 months
  Exercise capacity by VO2max test and/or submax test
Physical functioning | baseline, 12 weeks, 6 months and 15 months
  skeletal muscle strength by maximal strenght test
Body composition | baseline, 12 weeks, 6 months and 15 months
  waist circumference
Body composition | baseline, 12 weeks, 6 months and 15 months
  body fat percentage (bioelectrical impedance)
Body composition | baseline, 12 weeks, 6 months and 15 months
  Height and weight to calculate BMI
Cardiometabolic risk factors | baseline, 12 weeks, 6 months and 15 months
  Blood pressure
Cardiometabolic risk factors | baseline, 12 weeks, 6 months and 15 months
  Lipid profiles (cholesterol)
Cardiometabolic risk factors | baseline, 12 weeks, 6 months and 15 months
  Lipid profiles (triglycerides)
Cardiometabolic risk factors | baseline, 12 weeks and 15 months
  glucose metabolism
nutrition | baseline, 12 weeks, (6 months for nutrition intervention only) and 15 months
  dietary intake (food diaries)
nutrition | baseline and 15 months
  nutritional knowledge (questionnaire)
Psychological factors | 12 weeks and 15 months
  motivation (questionnaire)
Psychological factors | baseline and 15 months
  kinesiophobia (questionnaire)
Psychological factors | baseline
  coping style (questionnaire)
Chronic fatigue | baseline, 12 weeks, 6 months and 15 months
  CIS-20 questionnaire
Fatigue and work participation | baseline, 12 weeks, 6 months and 15 months
  Fatigue and work questionnaire (NFR)
Cost-effectiveness | baseline, 12 weeks, 6, 9, 12 and 15 months
  care consumption and intervention costs

CONTACTS AND LOCATIONS:
Overall Officials: Eva Corpleleijn, dr, Principal Investigator — University Medical Center Groningen
Locations (5):
- Netherlands (5):
  - Reade, Amsterdam, North Holland
  - Revalidatiecentrum Lindenhof, Goes, Zeeland
  - AMC, Amsterdam
  - Isala Kliniek, Zwolle
  - Vogellanden, Zwolle

REFERENCES:
- [Background] van den Ham EC, Kooman JP, Schols AM, Nieman FH, Does JD, Akkermans MA, Janssen PP, Gosker HR, Ward KA, MacDonald JH, Christiaans MH, Leunissen KM, van Hooff JP. The functional, metabolic, and anabolic responses to exercise training in renal transplant and hemodialysis patients. Transplantation. 2007 Apr 27;83(8):1059-68. doi: 10.1097/01.tp.0000259552.55689.fd. PMID 17452896
- [Background] van den Ham EC, Kooman JP, Schols AM, Nieman FH, Does JD, Franssen FM, Akkermans MA, Janssen PP, van Hooff JP. Similarities in skeletal muscle strength and exercise capacity between renal transplant and hemodialysis patients. Am J Transplant. 2005 Aug;5(8):1957-65. doi: 10.1111/j.1600-6143.2005.00944.x. PMID 15996245
- [Background] van den Ham EC. Body composition and exercise intolerance in renal transplant patients: the response to exercise training. Thesis. 2006.
- [Background] van den Ham EC, Kooman JP, Christiaans MH, Nieman FH, van Hooff JP. Weight changes after renal transplantation: a comparison between patients on 5-mg maintenance steroid therapy and those on steroid-free immunosuppressive therapy. Transpl Int. 2003 May;16(5):300-6. doi: 10.1007/s00147-002-0502-1. Epub 2003 Feb 20. PMID 12759720
- [Background] van den Ham EC, Kooman JP, Christiaans ML, van Hooff JP. The influence of early steroid withdrawal on body composition and bone mineral density in renal transplantation patients. Transpl Int. 2003 Feb;16(2):82-7. doi: 10.1007/s00147-002-0488-8. Epub 2003 Jan 18. PMID 12595969
- [Background] van den Ham EC, Kooman JP, Christiaans MH, Leunissen KM, van Hooff JP. Posttransplantation weight gain is predominantly due to an increase in body fat mass. Transplantation. 2000 Jul 15;70(1):241-2. No abstract available. PMID 10919614
- [Background] van den Ham EC, Kooman JP, Christiaans MH, van Hooff JP. Relation between steroid dose, body composition and physical activity in renal transplant patients. Transplantation. 2000 Apr 27;69(8):1591-8. doi: 10.1097/00007890-200004270-00013. PMID 10836368
- [Background] Zelle DM, Kok T, Dontje ML, Danchell EI, Navis G, van Son WJ, Bakker SJ, Corpeleijn E. The role of diet and physical activity in post-transplant weight gain after renal transplantation. Clin Transplant. 2013 Jul-Aug;27(4):E484-90. doi: 10.1111/ctr.12149. Epub 2013 Jun 13. PMID 23758229
- [Background] Zelle DM, Corpeleijn E, Stolk RP, de Greef MH, Gans RO, van der Heide JJ, Navis G, Bakker SJ. Low physical activity and risk of cardiovascular and all-cause mortality in renal transplant recipients. Clin J Am Soc Nephrol. 2011 Apr;6(4):898-905. doi: 10.2215/CJN.03340410. Epub 2011 Mar 3. PMID 21372213
- [Background] Kwakernaak AJ, Zelle DM, Bakker SJ, Navis G. Central body fat distribution associates with unfavorable renal hemodynamics independent of body mass index. J Am Soc Nephrol. 2013 May;24(6):987-94. doi: 10.1681/ASN.2012050460. Epub 2013 Apr 11. PMID 23578944
- [Background] Zelle DM, Corpeleijn E, Deinum J, Stolk RP, Gans RO, Navis G, Bakker SJ. Pancreatic beta-cell dysfunction and risk of new-onset diabetes after kidney transplantation. Diabetes Care. 2013 Jul;36(7):1926-32. doi: 10.2337/dc12-1894. Epub 2013 Feb 1. PMID 23378624
- [Background] Corpeleijn E, Bakker SJ, Stolk RP. Obesity and impaired renal function: potential for lifestyle intervention? Eur J Epidemiol. 2009;24(6):275-80. doi: 10.1007/s10654-009-9345-8. Epub 2009 May 7. PMID 19455406
- [Background] Mensink M, Corpeleijn E, Feskens EJ, Kruijshoop M, Saris WH, de Bruin TW, Blaak EE. Study on lifestyle-intervention and impaired glucose tolerance Maastricht (SLIM): design and screening results. Diabetes Res Clin Pract. 2003 Jul;61(1):49-58. doi: 10.1016/s0168-8227(03)00067-6. PMID 12849923
- [Background] Oterdoom LH, de Vries AP, Gansevoort RT, van Son WJ, van der Heide JJ, Ploeg RJ, de Jong PE, Gans RO, Bakker SJ. Determinants of insulin resistance in renal transplant recipients. Transplantation. 2007 Jan 15;83(1):29-35. doi: 10.1097/01.tp.0000245844.27683.48. PMID 17220787
- [Background] de Vries AP, Bakker SJ, van Son WJ, van der Heide JJ, Ploeg RJ, The HT, de Jong PE, Gans RO. Metabolic syndrome is associated with impaired long-term renal allograft function; not all component criteria contribute equally. Am J Transplant. 2004 Oct;4(10):1675-83. doi: 10.1111/j.1600-6143.2004.00558.x. PMID 15367224
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Hessels AC, van der Hoeven JH, Sanders JSF, Brouwer E, Rutgers A, Stegeman CA. Leg muscle strength is reduced and is associated with physical quality of life in Antineutrophil cytoplasmic antibody-associated vasculitis. PLoS One. 2019 Feb 4;14(2):e0211895. doi: 10.1371/journal.pone.0211895. eCollection 2019. PMID 30716132
- [Derived] Klaassen G, Zelle DM, Navis GJ, Dijkema D, Bemelman FJ, Bakker SJL, Corpeleijn E. Lifestyle intervention to improve quality of life and prevent weight gain after renal transplantation: Design of the Active Care after Transplantation (ACT) randomized controlled trial. BMC Nephrol. 2017 Sep 15;18(1):296. doi: 10.1186/s12882-017-0709-0. PMID 28915863